CLINICAL TRIAL: NCT04270279
Title: Efficacy and Safety of Xueshuanxinmaining Tablet for the Treatment of Stable Angina Pectoris: Multicenter, Randomised, Double Blind, Placebo Controlled Trial
Brief Title: Efficacy and Safety of Xueshuanxinmaining Tablet for the Treatment of Stable Angina Pectoris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun Li, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XSXMN_2019001
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Coronary Heart Disease; Stable Angina
Keywords: Coronary heart disease; Stable angina; Traditional Chinese medicine; Xueshuanxinmaining tablet
MeSH Terms: conditions — Coronary Disease; Angina, Stable | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xueshuanxinmaining Tablet (Experimental): Patients were given Xueshuanxinmaining tablet orally 2 pills each time, 3 times daily for 8 weeks. And patients can take nitroglycerin tablets provided by the sponsor when angina attack.
  For patients who have used drugs such as aspirin, angiotensin-converting enzyme inhibitor, lipid-lowering drugs to treat coronary heart disease before inclusion, they can continue to use the original varieties and doses, without dose adjustment.
  Interventions: Drug: Xueshuanxinmaining tablet; Drug: Nitroglycerin tablets
- Placebo (Placebo Comparator): Patients were given Xueshuanxinmaining tablet simulation orally 2 pills each time, 3 times daily for 8 weeks. And patients can take nitroglycerin tablets provided by the sponsor when angina attack.
  For patients who have used drugs such as aspirin, angiotensin-converting enzyme inhibitor, lipid-lowering drugs to treat coronary heart disease before inclusion, they can continue to use the original varieties and doses, without dose adjustment.
  Interventions: Drug: Xueshuanxinmaining placebo; Drug: Nitroglycerin tablets

INTERVENTIONS:
Drug: Xueshuanxinmaining tablet — A kind of Chinese patent medicine
  Other Names: XSXMN
  Arms: Xueshuanxinmaining Tablet
Drug: Xueshuanxinmaining placebo — The simulant of Xueshuanxinmaining tablet
  Other Names: XSXMN placebo
  Arms: Placebo
Drug: Nitroglycerin tablets — Be used when angina attack

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel clinical trial in Chinese population with stable angina pectoris. The purpose is to determine the efficacy and safety of Xueshuanxinmaining tablet in the treatment of stable angina pectoris.

DETAILED DESCRIPTION:
Xueshuanxinmaining tablet is a Chinese patent medicine composed of Ligusticum chuanxiong, Salvia miltiorrhiza, borneol and Toad puff, etc. It has been widely used in cardiovascular diseases in China. Clinical application suggested that Xueshuanxinmaining tablet was safe and effective in the treatment of stable angina pectoris. However, it still needs to be further confirmed by high-quality, large sample randomized controlled trials. This randomized, double-blind, placebo-controlled clinical trial is to determine the efficacy and safety of Xueshuanxinmaining tablet in the treatment of stable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged between 40 and 75 years.
* Meet the diagnostic criteria of stable angina pectoris.
* Meet Chinese medicine syndrome differentiation of Qi-yin deficiency and blood stasis syndrome.
* Voluntarily participate and sign informed consent.

Exclusion Criteria:

* Patients were diagnosed as acute myocardial infarction, unstable angina, stable exertion angina and other heart diseases.
* Patients with poor control of hypertension and diabetes, severe cardiopulmonary insufficiency, severe arrhythmia (rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia, etc.), with a history of heart pacemaker or cerebrovascular disease within one year.
* Any of the following disease history or evidence was found in the screening period: severe cardiovascular or cerebrovascular diseases; active, recurrent peptic ulcer or other bleeding risk diseases; other serious diseases of digestive system; combined with malignant tumor, blood system disease, serious or progressive diseases of the other system; combined with mental diseases.
* Before screening, any laboratory inspection index meets the following standards: The results showed that Glutamic aspartate transaminase (AST) or alanine aminotransferase (ALT) were more than 1.5 times of the upper limit of normal value and serum creatinine (Cr) was more than 1.2 times of the upper limit of normal value.
* With a history of alcohol and drug abuse.
* Pregnant or lactating women.
* Patients who have participated in clinical trials of other drugs within 3 months before enrollment.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Stopping or reducing rate of antianginal drugs | Eight weeks after treatment
  Antianginal drugs include nitroglycerin tablet, compound Danshen dropping pill and Suxiao Jiuxin pill.

SECONDARY OUTCOMES:
Stopping or reducing rate of antianginal drugs | Two, four and eight weeks after treatment
  Antianginal drugs include nitroglycerin tablet, compound Danshen dropping pill and Suxiao Jiuxin pill.
Changes of electrocardiogram (ECG) | Four and eight weeks after treatment
  Mainly observe the ST segment and the change of T wave from the baseline
Changes of Seattle Angina Questionnaire scores (SAQ scores) | Four and eight weeks after treatment
  The SAQ regroups 19 items measuring five specific scales: physical limitations, anginal stability, anginal frequency, treatment satisfaction and disease perception targeting a specific disease and treatment group. higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences